CLINICAL TRIAL: NCT05901961
Title: A Study of Effectiveness and Safety of Whitfield's Solution, Zinc Oxide Nanoparticles Solution and the Combination of Whitfield's and Zinc Oxide Nanoparticles Solution for the Treatment of Fungal Feet Infection
Brief Title: Effectiveness and Safety of Whitfield's Solution, Zinc Oxide Nanoparticles Solution or Combination for the Treatment of Fungal Feet Infection
Acronym: WhitfieldZinc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Dermatological Society of Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si 742/2020
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Fungal Foot Infection
Keywords: Whitfield; Zinc oxide nanoparticles; Fungal foot infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whitfield solution (Active Comparator): The patient will receive 60 mL of Whitfield solution. They will be instructed to apply 0.5 mL of the solution to the lesion twice daily for a consecutive period of 8 weeks.
  Interventions: Drug: Whitfield solution
- Zinc oxide nanoparticles solution (Active Comparator): The patient will receive 60 mL of 1% Zinc oxide nanoparticles solution. They will be instructed to apply 0.5 mL of the solution to the lesion twice daily for a consecutive period of 8 weeks.
  Interventions: Drug: Zinc oxide nanoparticles solution
- Combined Whitfield and Zinc oxide nanoparticles solution (Active Comparator): The patient will receive 60 mL of combined Whitfield and 1% Zinc oxide nanoparticles solution. They will be instructed to apply 0.5 mL of the solution to the lesion twice daily for a consecutive period of 8 weeks.
  Interventions: Drug: Combined Whitfield and Zinc oxide nanoparticles solution

INTERVENTIONS:
Drug: Whitfield solution — The patient will receive 60 mL of Whitfield solution. They will be instructed to apply 0.5 mL of the solution to the lesion twice daily for a consecutive period of 8 weeks.
  Arms: Whitfield solution
Drug: Zinc oxide nanoparticles solution — The patient will receive 60 mL of 1% Zinc oxide nanoparticles solution. They will be instructed to apply 0.5 mL of the solution to the lesion twice daily for a consecutive period of 8 weeks.
  Arms: Zinc oxide nanoparticles solution
Drug: Combined Whitfield and Zinc oxide nanoparticles solution — The patient will receive 60 mL of combined Whitfield and Zinc oxide nanoparticles solution. They will be instructed to apply 0.5 mL of the solution to the lesion twice daily for a consecutive period of 8 weeks.
  Arms: Combined Whitfield and Zinc oxide nanoparticles solution

SUMMARY:
This study aimed to study the efficacy of Whitfield's solution, zinc oxide nanoparticles solution, and the combination of Whitfield's and zinc oxide nanoparticles solution in treating fungal feet infection.

DETAILED DESCRIPTION:
Fungal foot infections are a common problem in medical practice, particularly among the elderly population. These infections can present in various ways, often characterized by dry and flaky skin on the feet. While the symptoms of fungal foot infections are generally gradual or even asymptomatic, they can lead to more severe complications, such as bacterial infections.

Topical antifungal drugs are primarily used for treating fungal foot infections, especially when the infection is localized and not present in other areas of the body. These medications have proven to be effective against dermatophyte fungal foot infections. However, in Thailand, fungal foot infections are frequently caused by non-dermatophyte species, which typically do not respond well to antifungal drugs. In such cases, topical peeling ointments like Whitfield Ointment are employed, as they offer favorable treatment outcomes for both dermatophyte and non-dermatophyte fungal foot infections. One drawback of Whitfield Ointment is its sticky consistency, which can adhere to surfaces, leading to irregular medication use by patients. At Siriraj Hospital, a Whitfield solution has been developed, although its therapeutic efficacy has yet to be studied. Nevertheless, based on its ingredients, it is expected to be similar to the ointment formulation.

Zinc oxide nanoparticles have exhibited activity against various bacteria and fungi, while remaining safe for human cells. They do not cause skin irritation and are not absorbed into the epidermis.

Based on a literature review, the use of zinc oxide nanoparticle solution and Whitfield solution for treating fungal foot infections has not been investigated. Therefore, our objective is to evaluate the effectiveness of zinc oxide nanoparticle solution alone, Whitfield solution alone, and a combination of Whitfield solution and zinc oxide nanoparticles in the treatment of fungal foot infections. Additionally, we aim to examine any potential side effects and assess user satisfaction with these treatments.

ELIGIBILITY:
Inclusion Criteria:

* The patient was diagnosed with a fungal foot infection based on the clinical presentation and a positive result from a microscopic examination for fungus.
* The patient must not have received any prior antifungal therapy, including topical, oral, or intravenous routes, within 36 weeks prior to recruitment.

Exclusion Criteria:

* Patients with conditions other than fungal foot infections, such as bacterial infections or inflammation of the skin on the foot
* Patients with other fungal diseases that require treatment with systemic antifungals, such as onychomycosis or tinea capitis
* Patients who are currently taking immunosuppressants or are immunocompromised.
* Patients who have difficulty applying the medication by themselves.
* Patients who have been treated for fungal foot infection using methods that are not included in the research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2023-09-09 (Actual)

PRIMARY OUTCOMES:
Efficacy between Whitfield solution, zinc oxide nanoparticles particle, and a combination of Whitfield and Zinc oxide nanoparticles in treating fungal foot infection. | 4 weeks and 8 weeks
  The efficacy of Whitfield solution, zinc oxide nanoparticles, and a combination of Whitfield solution and zinc oxide nanoparticles in treating fungal foot infections will be evaluated by comparing the proportion of patients with negative results from the KOH test for fungal infection at both 4 weeks and 8 weeks.

SECONDARY OUTCOMES:
Safety between Whitfield solution, zinc oxide nanoparticles particle, and a combination of Whitfield and Zinc oxide nanoparticles in treating fungal foot infection. | 4 weeks and 8 weeks
  The safety of Whitfield solution, zinc oxide nanoparticles, and a combination of Whitfield solution and zinc oxide nanoparticles in treating fungal foot infections will be evaluated by comparing the incidence of adverse effects resulting from each medication in each group at both 4 weeks and 8 weeks.
Comparing patients' satisfaction between using Whitfield solution, zinc oxide nanoparticles particle, and a combination of Whitfield and Zinc oxide nanoparticles in treating fungal foot infection. | 4 weeks and 8 weeks
  The satisfaction of patients using Whitfield solution, zinc oxide nanoparticles, and a combination of Whitfield solution and zinc oxide nanoparticles in treating fungal foot infections will be evaluated at both 4 weeks and 8 weeks by asking the patients to rate their satisfaction score on the 5-point Likert scale from 0 to 4 (Higher scores mean a a better outcome).
The diversity of microbiome in fungal foot infection patients before and 8 weeks after treatment | 8 weeks
  The composition of the microbiome in patients with fungal foot infections will be evaluated before and 8 weeks after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Charussri Leeyaphan, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Dermatology Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gooskens V, Ponnighaus JM, Clayton Y, Mkandawire P, Sterne JA. Treatment of superficial mycoses in the tropics: Whitfield's ointment versus clotrimazole. Int J Dermatol. 1994 Oct;33(10):738-42. doi: 10.1111/j.1365-4362.1994.tb01524.x. PMID 8002148
- [Background] WILLIAMS DI. The Whitfield tradition of therapy. Br Med J. 1955 Aug 20;2(4937):453-5. doi: 10.1136/bmj.2.4937.453. No abstract available. PMID 13240146
- [Background] Gondal MA, Alzahrani AJ, Randhawa MA, Siddiqui MN. Morphology and antifungal effect of nano-ZnO and nano-Pd-doped nano-ZnO against Aspergillus and Candida. J Environ Sci Health A Tox Hazard Subst Environ Eng. 2012;47(10):1413-8. doi: 10.1080/10934529.2012.672384. PMID 22571529
- [Background] Krol A, Pomastowski P, Rafinska K, Railean-Plugaru V, Buszewski B. Zinc oxide nanoparticles: Synthesis, antiseptic activity and toxicity mechanism. Adv Colloid Interface Sci. 2017 Nov;249:37-52. doi: 10.1016/j.cis.2017.07.033. Epub 2017 Aug 26. PMID 28923702
- [Background] Mihai MM, Dima MB, Dima B, Holban AM. Nanomaterials for Wound Healing and Infection Control. Materials (Basel). 2019 Jul 6;12(13):2176. doi: 10.3390/ma12132176. PMID 31284587
- [Background] Vinardell MP, Llanas H, Marics L, Mitjans M. In Vitro Comparative Skin Irritation Induced by Nano and Non-Nano Zinc Oxide. Nanomaterials (Basel). 2017 Mar 4;7(3):56. doi: 10.3390/nano7030056. PMID 28336890
- [Background] Leite-Silva VR, Sanchez WY, Studier H, Liu DC, Mohammed YH, Holmes AM, Ryan EM, Haridass IN, Chandrasekaran NC, Becker W, Grice JE, Benson HA, Roberts MS. Human skin penetration and local effects of topical nano zinc oxide after occlusion and barrier impairment. Eur J Pharm Biopharm. 2016 Jul;104:140-7. doi: 10.1016/j.ejpb.2016.04.022. Epub 2016 Apr 27. PMID 27131753
- [Background] Tiwari N, Pandit R, Gaikwad S, Gade A, Rai M. Biosynthesis of zinc oxide nanoparticles by petals extract of Rosa indica L., its formulation as nail paint and evaluation of antifungal activity against fungi causing onychomycosis. IET Nanobiotechnol. 2017 Mar;11(2):205-211. doi: 10.1049/iet-nbt.2016.0003. PMID 28477005
- [Result] Vander Straten MR, Hossain MA, Ghannoum MA. Cutaneous infections dermatophytosis, onychomycosis, and tinea versicolor. Infect Dis Clin North Am. 2003 Mar;17(1):87-112. doi: 10.1016/s0891-5520(02)00065-x. PMID 12751262
- [Result] 2. Nigam PK, Saleh D. Tinea Pedis. [Updated 2020 May 3]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing. Available from: https://www.ncbi.nlm.nih.gov/books/NBK470421/. Accessed August 22, 2020.
- [Derived] Leeyaphan C, Punnakitikashem P, Suiwongsa B, Komesmuneeborirak P, Chongtrakool P, Kulthanachairojana N, Limphoka P, Hutachoke T, Saengthong-Aram P, Kobkurkul P, Wongdama S, Pongkittilar B, Matthapan L, Panyawong C, Prasong W, Plengpanich A, Kunwong N, Rodponthukwaji K, Bunyaratavej S. Efficacy, Safety, and Cost-effectiveness of Zinc Oxide Nanoparticles in Whitfield's Spirit Solution for Treating Superficial Fungal Foot Infections: A Randomized Controlled Trial. Dermatol Ther (Heidelb). 2025 Feb;15(2):351-365. doi: 10.1007/s13555-025-01340-2. Epub 2025 Jan 27. PMID 39871011